CLINICAL TRIAL: NCT05127811
Title: A Phase I Dose Escalation Study of ZN-d5 Monotherapy in Chinese Subjects With Non-Hodgkin Lymphoma
Brief Title: A Phase I Study of ZN-d5 in Chinese Subjects With Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Zentera Therapeutics HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: d5ZTCN100
Record Dates: First submitted 2021-09-18; First posted 2021-11-19 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- 100mg(on empty) (Experimental)
  Interventions: Drug: ZN-d5
- 200mg(on empty) (Experimental)
  Interventions: Drug: ZN-d5
- 400mg(on empty) (Experimental)
  Interventions: Drug: ZN-d5
- 600mg(on empty) (Experimental)
  Interventions: Drug: ZN-d5
- 600mg（with a meal） (Experimental)
  Interventions: Drug: ZN-d5
- 800mg(with a meal) (Experimental)
  Interventions: Drug: ZN-d5

INTERVENTIONS:
Drug: ZN-d5 — BION design

SUMMARY:
A phase I dose-escalation, open-label, multicenter study to assess the safety, tolerability, clinical activity, and pharmacokinetics (PK) of ZN-d5 in Chinese subjects with non-Hodgkin lymphoma (NHL).

DETAILED DESCRIPTION:
For the Phase I dose escalation study of ZN-d5, it is planned that after the starting dose, subsequent dose assignments will be made by means of a model-assisted design, until the MTD or RP2D is determined in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. NHL, relapsed from or refractory to at least 2 prior lines of systemic therapy (excluding radiotherapy and surgery); subjects must have failed or not be candidates for available standard therapy expected to provide clinical benefit.
2. Female subjects of childbearing potential must have a negative serum pregnancy test and agree to use contraception while on study.
3. Eastern Cooperative Oncology Group performance status ≤ 1.
4. Adequate blood and other organ function, defined by the following criteria:

   1. Neutrophil count (ANC) ≥ 1.0 × 109/L.
   2. Platelet count ≥ 75 × 109/L at least 3 days after platelet transfusion (≥ 50 × 109/L permitted if the bone marrow is > 50% lymphoma cells).
   3. Hemoglobin ≥ 8.0 g/dL.
   4. Coagulation parameters ≤ 1.5 × upper limit of normal (ULN).
   5. Liver enzymes ≤ 3 × ULN and total bilirubin ≤ 1.5 × ULN.
   6. Creatinine clearance ≥ 60 mL/min.

Exclusion Criteria:

1. Received any of the following prior to start of ZN-d5 treatment:

   1. Systemic administration of antineoplastic agents (including investigational agents) within the shorter of 28 days or 5 half-lives.
   2. Major surgery within 28 days.
   3. Radiotherapy within 14 days.
   4. Autologous or allogeneic stem cell transplantation within 60 days, or receiving immunosuppression for active graft-versus-host disease.
   5. Use of strong CYP3A4 inhibitors, P-gp inhibitors or QT prolonging agents within 5 half-lives, or potent or moderate CYP3A4 inducers within 14 days.
2. Ongoing and clinically significant non-hematologic toxicity related to prior antineoplastic therapy.
3. Presence of major cardiovascular system diseases (including QTcF > 480 msec).
4. Positive serology for human immunodeficiency virus, hepatitis B, or hepatitis C unless no detectable hepatitis B or C viral load.
5. Unable to take oral drugs or presence of severe gastrointestinal abnormalities.
6. Active and uncontrolled clinically significant infection.
7. Other active systemic malignancy or other severe, unstable, or poorly controlled acute or chronic medical conditions.
8. Prior treatment with venetoclax or other BCL-2 inhibitors.
9. Primary or secondary CNS lymphoma.
10. Presence of post-transplant lymphoproliferative disease, Burkitt's lymphoma, Burkitt-like lymphoma, T lymphoblastic lymphoma and T lymphoblastic acute leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Safety monitoring | until 30 days after the last dose of study drug
  Incidence and severity of adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
DLT | at the end of Cycle 1
  Dose-limiting toxicities (DLTs) observed in DLT evaluable subjects

SECONDARY OUTCOMES:
Effacy Evaluation | up to 24 months
  Efficacy as defined by the 2014 Lugano response criteria
Maximum Plasma Concentration [Cmax] | up to 24 months
  Plasma PK parameters of ZN-d5

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - BeiJing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yan Set University Cancer Center, Guangzhou, Guangdong
  - Fudan University Shanghai Cancer Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided